CLINICAL TRIAL: NCT04322539
Title: A Global Multicenter Randomized Placebo-Controlled Phase 3 Trial To Compare The Efficacy And Safety Of Fruquintinib Plus Best Supportive Care To Placebo Plus Best Supportive Care In Patients With Refractory Metastatic Colorectal Cancer
Brief Title: A Study of Efficacy and Safety of Fruquintinib (HMPL-013) in Participants With Metastatic Colorectal Cancer
Acronym: FRESCO-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hutchison Medipharma Limited (Industry)
Responsible Party: Sponsor
Organization: Hutchmed (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019-013-GLOB1
Record Dates: First submitted 2020-03-24; First posted 2020-03-26 (Actual); Results first posted 2023-09-14 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Metastatic Colorectal Cancer; Metastatic Colon Cancer
Keywords: colon; colorectal; mcrc; crc; metastatic colon; metastatic colorectal; VEGF; VEGFR
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — HMPL-013

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fruquintinib Plus Best Supportive Care (BSC) Group (Experimental): Participants will be orally administered Fruquintinib 5 mg in combination with BSC once daily for 3 weeks of continuous dosing followed by a 1-week break (with each cycle length of 28 days).
  Interventions: Drug: Fruquintinib
- Placebo Plus BSC Group (Placebo Comparator): Participants will be orally administered Placebo 5 mg in combination with BSC once daily for 3 weeks of continuous dosing followed by a 1-week break (with each cycle length of 28 days).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fruquintinib — Oral VEGFR inhibitor
  Other Names: HMPL-013
  Arms: Fruquintinib Plus Best Supportive Care (BSC) Group
Drug: Placebo — Placebo capsule
  Arms: Placebo Plus BSC Group

SUMMARY:
This is a global, randomized, double-blind, placebo-controlled, multicenter phase 3 clinical trial to compare the efficacy and safety of fruquintinib plus best supportive care (BSC) versus placebo plus BSC in participants with refractory metastatic colorectal cancer (mCRC). 691 participants were randomized to one of the following treatment arms in a 2:1 ratio, fruquintinib plus BSC or placebo plus BSC.

DETAILED DESCRIPTION:
This is a global, randomized, double-blind, placebo-controlled, multicenter phase 3 clinical trial to compare the efficacy and safety of fruquintinib in combination with BSC versus placebo in combination with BSC in metastatic colorectal cancer participants who have progressed on, or were intolerant to, chemotherapy, anti-VEGF and anti-EGFR biologics, and TAS-102 or regorafenib. Participants with MSI-H/MMR deficient tumors must have also received an immune checkpoint inhibitor if approved and available and if deemed appropriate. Subjects with BRAF-mutant tumors must have been treated with a BRAF inhibitor if approved and available and if deemed appropriate.

Metastatic colorectal cancer cannot be cured by surgery. Therefore, treatment principals are primarily aimed at controlling disease progression and prolonging survival. Standard first- and second-line therapy includes cytotoxic drugs such as 5-fluorouracil, oxaliplatin, and irinotecan; anti-VEGF therapy; and, if RAS wild type, anti-EGFR therapy. After the first two lines of chemotherapy, standard third-line treatment is either TAS-102 or regorafenib. There are currently no effective treatments for patients who have progressed on standard, approved therapies, and treatment options include reuse of prior therapies, clinical trials or BSC. Consequently, there is an unmet medical need for additional safe and effective treatment.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent;
* Age ≥18 years;
* Histologically and/or cytologically documented metastatic colorectal adenocarcinoma. RAS, BRAF, and microsatellite instability microsatellite instability (MSI)/mismatch repair (MMR) status for each patient must be documented, according to country level guidelines;
* Participants must have progressed on or been intolerant to treatment with either trifluridine/tipiracil (TAS-102) or regorafenib. Participants are considered intolerant to TAS-102 or regorafenib if they have received at least 1 dose of either agents and were discontinued from therapy for reasons other than disease progression. Participants who have been treated with both TAS-102 and regorafenib are permitted. Participants must also have been previously treated with standard approved therapies: fluoropyrimidine-, oxaliplatin-, and irinotecan-based chemotherapy, an anti-VEGF biological therapy, and, if RAS wild-type, an anti-EGFR therapy;
* Participants with microsatellite-high (MSI-H) or mismatch repair deficient (dMMR) tumors must have been treated with immune checkpoint inhibitors if approved and available in the participant's country unless the patient is ineligible for treatment with a checkpoint inhibitor;
* Participants who received oxaliplatin in the adjuvant setting and developed metastatic disease during or within 6 months of completing adjuvant therapy are considered eligible without receiving oxaliplatin in the metastatic setting. Participants who developed metastatic disease more than 6 months after completion of oxaliplatin-containing adjuvant treatment must be treated with oxaliplatin-based therapy in the metastatic setting to be eligible;
* Body weight ≥40kg;
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1;
* Have measurable disease according to RECIST Version 1.1, assessed locally. Tumors that were treated with radiotherapy are not measurable per RECIST Version 1.1, unless there has been documented progression of those lesions;
* Expected survival >12 weeks.
* For female participants of childbearing potential and male participants with partners of childbearing potential, agreement to use a highly effective form(s) of contraception, that results in a low failure rate (<1% per year) when used consistently and correctly, starting during the screening period, continuing throughout the entire study period, and for 90 days after taking the last dose of study drug. Such methods include: oral hormonal contraception (combined estrogen/ progestogen, or progestogen-only) associated with inhibition of ovulation, intrauterine device (IUD), intrauterine hormone-releasing system (IUS), bilateral tubal ligation, vasectomized partner, or true sexual abstinence in line with the preferred and usual lifestyle of the participant. Highly effective contraception should always be combined with an additional barrier method (eg, diaphragm, with spermicide). The same criteria are applicable to male participants involved in this clinical trial if they have a partner of childbirth potential, and male participants must always use a condom.
* Participants with BRAF-mutant tumors must have been treated with a BRAF inhibitor if approved and available in the participant's home country unless the patient is ineligible for treatment with a BRAF inhibitor.

Exclusion Criteria:

* Absolute neutrophil count (ANC) <1.5×109/L, platelet count <100×109/L, or hemoglobin <9.0 g/dL. Blood transfusion within 1 week prior to enrollment for the purpose of increasing the likelihood of eligibility is not allowed;
* Serum total bilirubin >1.5 × the upper limit of normal (ULN). Participants with Gilbert syndrome, bilirubin <2 X ULN, and normal AST/ALT are eligible;
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2.5 × ULN in participants without hepatic metastases; ALT or AST >5 × ULN in participants with hepatic metastases;
* Serum creatinine >1.5 × ULN or creatinine clearance <60 mL/min. Creatinine clearance can either be measured in a 24-hour urine collection or estimated by the Cockroft-Gault equation.
* Urine dipstick protein ≥2+ or 24-hour urine protein ≥1.0 g/24-h. Participants with greater than 2+ proteinuria by dipstick must undergo a 24-hour urine collection to assess urine protein level;
* Uncontrolled hypertension, defined as: systolic blood pressure ≥140 mm Hg and/or diastolic blood pressure ≥90 mm Hg despite optimal medical management. Participants were required to have blood pressure values below both limits. Repeated assessments were permitted;
* International Normalized Ratio (INR) >1.5 x ULN or activated partial thromboplastin time (aPTT) >1.5 × ULN, unless the patient is currently receiving or intended to receive anticoagulants for prophylactic purposes;
* History of, or active gastric/duodenal ulcer or ulcerative colitis, active hemorrhage of an unresected gastrointestinal tumor, history of perforation or fistulas; or any other condition that could, in the investigator's judgment, result in gastrointestinal hemorrhage or perforation; within the 6 months prior to screening;
* History or presence of hemorrhage from any other site (eg, hemoptysis or hematemesis) within 2 months prior to screening;
* History of a thromboembolic event, including deep vein thrombosis (DVT), pulmonary embolism (PE), or arterial embolism within 6 months prior to screening.
* Stroke and/or transient ischemic attack within 12 months prior to screening;
* Clinically significant cardiovascular disease, including but not limited to acute myocardial infarction or coronary artery bypass surgery within 6 months prior to enrollment, severe or unstable angina pectoris, New York Heart Association Class III/IV congestive heart failure, ventricular arrhythmias requiring treatment, or left ventricular ejection fraction (LVEF) <50% by echocardiogram;
* Mean corrected QT interval using the Fridericia method (QTcF) >480 msec or any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as hypokalemia, congenital long QT syndrome, family history of long QT syndrome, or unexplained sudden death under 40 years of age in a first-degree relative.
* Concomitant medications with a known risk of causing QT prolongation and/or Torsades de Pointes.
* Systemic anti-neoplastic therapies (except for those described in Exclusion 18) or any investigational therapy within 4 weeks prior to the first dose of study drug, including chemotherapy, radical radiotherapy, hormonotherapy, biotherapy and immunotherapy;
* Systemic small molecule targeted therapies (eg, tyrosine kinase inhibitors) within 5 half-lives or 4 weeks (whichever is shorter) prior to the first dose of study drug;
* Palliative radiotherapy for bone metastasis/lesion within 2 weeks prior to the initiation of study drug;
* Brachytherapy (i.e., implantation of radioactive seeds) within 60 days prior to the first dose of study drug.
* Use of strong inducers or inhibitors of CYP3A4 within 2 weeks (or 5 half-lives, whichever is longer) before the first dose of study drug;
* Surgery or invasive procedure (i.e., a procedure that includes a biopsy; central venous catheter placement is allowed) within 60 days prior to the first dose of study drug or unhealed surgical incision;
* Any unresolved toxicities from a previous antitumor treatment greater than CTCAE v5.0 Grade 1 (except for alopecia or neurotoxicity grade≤2);
* Known human immunodeficiency virus (HIV) infection;
* Known history of active viral hepatitis. For participants with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated. Participants with HCV infection who are currently on treatment are eligible if they have an undetectable HCV viral load.
* Clinically uncontrolled active infection requiring IV antibiotics;
* Tumor invasion of a large vascular structure, eg, pulmonary artery, superior or inferior vena cava;
* Women who are pregnant or lactating;
* Brain metastases and/or spinal cord compression untreated with surgery and/or radiotherapy, and without clinical imaging evidence of stable disease for 14 days or longer; participants requiring steroids within 4 weeks prior to start of study treatment are excluded;
* Other malignancy, except for non-melanoma skin cancer, in situ cervical ca or bladder ca (Tis and T1) that have been adequately treated during the 5 years prior to screening;
* Inability to take medication orally, dysphagia or an active gastric ulcer resulting from previous surgery (eg, gastric bypass) or a severe gastrointestinal disease, or any other condition that investigators believe may affect absorption of the investigational product;
* Other disease, metabolic disorder, physical examination anomaly, abnormal laboratory result, or any other condition (e.g., current alcohol or drug abuse) that investigators suspect may prohibit use of the investigational product, affect interpretation of study results, or put the patient at undue risk of harm based on the investigator's assessment;
* Known hypersensitivity to fruquintinib (or placebo) or any of its inactive ingredients including the azo dyes Tartrazine - FD&C Yellow 5 and Sunset yellow FCF - FD&C Yellow 6;
* Participants who have received prior fruquintinib;
* Live vaccine <28days before the first dose of study drug(s). Seasonal vaccines for influenza are generally inactivated vaccines and are allowed. Intranasal vaccines are live vaccines and are not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 691 (Actual)
Dates: Start 2020-08-12 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2024-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Schelman, MD, PhD, Study Director — HUTCHMED International Corporation
Locations (153):
- United States (45):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Arizona Oncology Associates, PC-HOPE, Tucson, Arizona
  - California Research Institute (CRI), Los Angeles, California
  - City of Hope Comprehensive Cancer Center, Los Angeles, California
  - Rocky Mountain Cancer Center, Aurora, Colorado
  - The George Washington University Medical Center, Washington D.C., District of Columbia
  - Sarah Cannon Research Institute-S-Ft. Myers (FCS South), Fort Myers, Florida
  - Mayo Clinic Florida, Jacksonville, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Cancer Care Centers of Brevard, Inc., Palm Bay, Florida
  - Sarah Cannon Research Institute-N-St Pete (FCS North), St. Petersburg, Florida
  - Sarah Cannon Research Institute-Pan-Tallahassee (FCS Panhandle), Tallahassee, Florida
  - Sarah Cannon Research-E-WPB (Florida Cancer Specialists-FCS East), West Palm Beach, Florida
  - Emory Winship Cancer Institute, Atlanta, Georgia
  - Illinois Cancer Specialists, Arlington Heights, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Affiliated Oncologists, Chicago Ridge, Illinois
  - XCancer / Central Care Cancer Center, Garden City, Kansas
  - University of Louisville - James Brown Cancer Center, Louisville, Kentucky
  - Norton Cancer Institute Audubon, Louisville, Kentucky
  - Hematology Oncology Clinic, Baton Rouge, Louisiana
  - XCancer / Pontchartrain Cancer Center, Hammond, Louisiana
  - Maryland Oncology Hematology, P.A., Columbia, Maryland
  - University of Michigan Health System, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Minnesota Oncology, Minneapolis, Minnesota
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Center for Pharmaceutical Research, Kansas City, Missouri
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - XCancer / New Mexico Oncology & Hematology Consultants, Albuquerque, New Mexico
  - Charleston Oncology, Charleston, South Carolina
  - Sarah Cannon Tennessee Oncology, Nashville, Tennessee
  - Vanderbilt Ingram Cancer Center, Nashville, Tennessee
  - Texas Oncology - Austin, Austin, Texas
  - Texas Oncology Baylor Sammons, Dallas, Texas
  - Texas Oncology-El Paso, El Paso, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Texas Oncology-McAllen, McAllen, Texas
  - Texas Oncology-San Antonio, San Antonio, Texas
  - Texas Oncology-Tyler, Tyler, Texas
  - Virginia Oncology Associates, Norfolk, Virginia
  - Providence Regional Cancer Partnership, Everett, Washington
  - Northwest Cancer Specialists, P.C., Vancouver, Washington
  - Medical College of Wisconsin/ Froedtert Hospital, Milwaukee, Wisconsin
- Australia (6):
  - Integrated Clinical Oncology Network Pty Ltd (Icon), Brisbane, Queensland
  - The Queen Elizabeth Hospital, Adelaide, South Australia
  - Flinders Medical Centre, Adelaide, South Australia
  - Western Health, Melbourne, Victoria
  - Austin Hopistal Medical Oncology Unit, Melbourne, Victoria
  - Monash Health, Melbourne, Victoria
- Austria (6):
  - Ordensklinikum Linz Barmherzige Schwestern, Linz, AUT
  - Schwerpunktkrankenhaus Feldkirch, Rankweil, AUT
  - Klinikum Steyr, Steyr, AUT
  - Wiener Gesundheitsverbund - Klinik Ottakring, Vienna, AUT
  - Klinikum Wels-Grieskirchen GmbH, Wels, AUT
  - Landesklinikum Wiener Neustadt, Wiener Neustadt, AUT
- Belgium (11):
  - Onze-Lieve-Vrouwziekenhuis OLV - Campus Aalst, Aalst, BEL
  - UCL St-Luc, Brussels, BEL
  - Grand Hopital de Charleroi, Charleroi, BEL
  - UZ Antwerpen, Edegem, BEL
  - Centres Hospitaliers Jolimont, Haine-Saint-Paul, BEL
  - UZ Leuven, Leuven, BEL
  - AZ Delta Roeselare, Roeselare, BEL
  - AZ Turnhout, Turnhout, BEL
  - CHU Mont-Godinne, Yvoir, BEL
  - Clinique CHC MontLegia, Liège, Wallonia
  - CHU de Lige - Domaine Universitaire du Sart Tilman, Liège, Wallonia
- Czechia (3):
  - Masaryk Memorial Cancer Institute, Hematoonkologie, Brno, Moravia
  - Fakultni nemocnice Olomouc, Onkologicka klinika, Olomouc, Moravia
  - Vseobecna Fakultni Nemocnice VFN, Onkologicka Klinika, Prague
- Estonia (3):
  - East Tallinn Central Hospital Centre of Oncology, Tallinn, Harju
  - Sihtasutus Pohja-Eesti Regionaalhaigla (PERH) (North Estonia Medical Centre), Tallinn, Harju
  - Tartu University Hospital Clinic of Haematology and Oncology, Tartu
- France (13):
  - CHU Besancon, Besançon, Franche-Comte
  - Institut Bergonie, Bordeaux, FRA
  - Unicancer, Caen, FRA
  - Centre Georges-Francois Leclerc, Dijon, FRA
  - ICM-Val d'Aurelle, Montpellier, FRA
  - Saint-Louis Hospital, Paris, FRA
  - Hopital St Antoine, Paris, FRA
  - Hopital Pitie Salptriere, Paris, FRA
  - CHU Poitiers, Poitiers, FRA
  - Centre hospitalier Annecy Genevois, Pringy, FRA
  - Centre Hospitalier Universitaire CHU de Rennes - Hopital de Pontchaillou, Rennes, FRA
  - Institut de cancerologie Strasbourg-Europe, Strasbourg, FRA
  - Institut Gustave Roussy, Villejuif, Paris
- Germany (13):
  - Universitaetsklinikum Erlangen, Erlangen, Bavaria
  - HELIOS Klinikum Berlin-Buch Saarow, Berlin, DEU
  - Charite - Universitaetsmedizin Berlin, Berlin, DEU
  - Universitaetsklinik Dresden, Dresden, DEU
  - University Hospital Essen, Essen, DEU
  - Institut fr Klinisch Onkologische ForschungKrankenhaus Nordwest GmbH, Frankfurt am Main, DEU
  - Haematologisch-Onkologische Praxis Hamburg Eppendorf, Hamburg, DEU
  - Asklepios Tumorzentrum Hamburg AK Altona, Hamburg, DEU
  - Universitaeres Krebszentrum Leipzig, Leipzig, DEU
  - RKH Kliniken, Ludwigsburg, DEU
  - Universitaetsmedizin Mannheim- III. Medizinische Klinik, Mannheim, DEU
  - Klinikum Neuperlach, München, DEU
  - Zentrum für Hämatologie und Onkologie MVZ GmbH, Porta Westfalica, DEU
- Hungary (11):
  - Del-Pesti Centrumkorhaz Orszagos Hematologiai es Infektologiai Intezet, Szent Laszlo Korhaz, Budapest, HUN
  - National Institute of Oncology, Budapest, HUN
  - Magyar Honvedseg Egeszsegugyi Kozpont, Budapest, HUN
  - Debreceni Egyetem Klinikai Kozpont, Debrecen, HUN
  - Bacs- Kiskun Megyei Korhaz, Kecskemét, HUN
  - Szabolcs-Szatmar-Bereg megyei Korhazak es Egyetemi Oktatokorhaz, Nyíregyháza, HUN
  - Hetenyi G Korhaz, Onkologiai Kozpont, Szolnok, HUN
  - Szent Borbala Korhaz, Tatabánya, HUN
  - Somogy Megyei Kaposi Mor Oktato Korhaz, Klinikai Onkologiai Osztaly, Kaposvár, Somogy County
  - Zala Megyei Szent Rafael Korhaz, Onkologiai Osztaly, F epulet 3. em., Zalaegerszeg, Zala County
  - Bekes Megyei Kozponti Korhaz, Pandy Kalman Tagkorhaz, Megyei Onkologiai Kozpont, Gyula
- Italy (11):
  - Fondazione Poliambulanza Hospital, Brescia, ITA
  - Policlinico San Martino di Genova, Genova, ITA
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, ITA
  - ASST Grande Ospedale Metropolitano Niguarda, Milan, ITA
  - Istituto Nazionale Tumori IRCCS Fondazione G. Pascale, Naples, ITA
  - Istituto Oncologico Veneto Irccs, Padua, ITA
  - Azienda Ospedaliero Universitaria Pisana, Pisa, ITA
  - Azienda USL-IRCCS di Reggio Emilia, Reggio Emilia, ITA
  - AO Card G Panico, Tricase, ITA
  - Ospedale San Bortolo Azienda ULSS8 Berica - Distretto Est, Vicenza, ITA
  - Istituto Clinico Humanitas, Rozzano MI, Lombardy
- Japan (10):
  - Aichi Cancer Center, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - Shikoku Cancer Center, Matsuyama, Ehime
  - Kyushu Cancer Center, Fukuoka, Fukuoka
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - St. Marianna University School of Medicine Hospital, Kawasaki-shi, Kanagawa
  - Kindai University Hospital, Osakasayama-shi, Osaka
  - Osaka University Hospital, Suita-shi, Osaka
  - Shizuoka Cancer Center, Shizuoka, Sunto-gun
  - National Cancer Center Hospital, Chuo-ku, Tokyo
- Poland (2):
  - M Sklodowska Curie Memorial Cancer Center, Klinika Gastroenterologii Onkologicznej, Warsaw, Masovia
  - Bialostockie Centrum Onkologii im. Marii Skodowskiej-Curie, Bialystok, Podlaskie Voivodeship
- Spain (16):
  - Hospital Universitari Vall dHebron, Barcelona, ESP
  - Hospital Universitario Reina Sofa, Córdoba, ESP
  - Hospital General Universitario de Elche, Elche, ESP
  - Hospital Universitario Ramón y Cajal, Madrid, ESP
  - Hospital Clinico San Carlos, Madrid, ESP
  - Hospital Universitario 12 de Octubre, Madrid, ESP
  - Hospital Universitario La Paz, Madrid, ESP
  - Hospital Universitario HM Sanchinarro, Madrid, ESP
  - Hospital Universitario Puerta de Hierro, Majadahonda, ESP
  - Hospital Regional Universitario Carlos Haya, Málaga, ESP
  - Hospital Universitario Central de Asturias, Oviedo, ESP
  - Hospital Universitario Marques de Valdecilla, Santander, ESP
  - Hospital ClÃ-nico Universitario de Santiago-CHUS, Santiago de Compostela, ESP
  - Hospital General Universitario Gregorio Maranon HGUGM, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Clinico Universitario de Valencia, Valencia
- United Kingdom (3):
  - Aberdeen Royal Infirmary, Aberdeen, GBR
  - The Royal Marsden Hospital, London, GBR
  - Sarah Cannon Research Institute UK, London, Middlesex

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kotani D, Yoshino T, Masuishi T, Sunakawa Y, Takashima A, Yamazaki K, Kawakami H, Nishina T, Komatsu Y, Esaki T, Eng C, Ukrainskyj S, Pallai R, Nanda S, Yang Z, Schelman W, Kania M, Satoh T. Efficacy and safety of fruquintinib in patients with refractory metastatic colorectal cancer: a FRESCO-2 subgroup analysis of patients enrolled in Japan. Int J Clin Oncol. 2025 Oct;30(10):2043-2052. doi: 10.1007/s10147-025-02852-9. Epub 2025 Sep 1. PMID 40888992
- [Derived] Sobrero A, Dasari A, Aquino J, Lonardi S, Garcia-Carbonero R, Elez E, Yoshino T, Yao J, Garcia-Alfonso P, Kocsis J, Gracian AC, Sartore-Bianchi A, Satoh T, Randrian V, Tomasek J, Chong G, Price T, Yu Z, Geiger A, Chen L, Yang Z, Schelman WR, Kania M, Tabernero J, Eng C. Health-related quality of life associated with fruquintinib in patients with metastatic colorectal cancer: Results from the FRESCO-2 study. Eur J Cancer. 2025 Mar 11;218:115268. doi: 10.1016/j.ejca.2025.115268. Epub 2025 Jan 29. PMID 39952149
- [Derived] Dasari A, Lonardi S, Garcia-Carbonero R, Elez E, Yoshino T, Sobrero A, Yao J, Garcia-Alfonso P, Kocsis J, Cubillo Gracian A, Sartore-Bianchi A, Satoh T, Randrian V, Tomasek J, Chong G, Paulson AS, Masuishi T, Jones J, Csoszi T, Cremolini C, Ghiringhelli F, Shergill A, Hochster HS, Krauss J, Bassam A, Ducreux M, Elme A, Faugeras L, Kasper S, Van Cutsem E, Arnold D, Nanda S, Yang Z, Schelman WR, Kania M, Tabernero J, Eng C; FRESCO-2 Study Investigators. Fruquintinib versus placebo in patients with refractory metastatic colorectal cancer (FRESCO-2): an international, multicentre, randomised, double-blind, phase 3 study. Lancet. 2023 Jul 1;402(10395):41-53. doi: 10.1016/S0140-6736(23)00772-9. Epub 2023 Jun 15. PMID 37331369
- [Derived] Dasari A, Sobrero A, Yao J, Yoshino T, Schelman W, Yang Z, Chien C, Kania M, Tabernero J, Eng C. FRESCO-2: a global Phase III study investigating the efficacy and safety of fruquintinib in metastatic colorectal cancer. Future Oncol. 2021 Aug;17(24):3151-3162. doi: 10.2217/fon-2021-0202. Epub 2021 May 17. PMID 33993740

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 124 study sites in the United States, Europe region, Japan, and Australia.
Pre-assignment Details: A total of 691 participants were randomized and enrolled in this study.
Groups:
- Fruquintinib + Best Supportive Care (BSC) Group: Participants received 5 milligrams (mg) of fruquintinib oral capsule in combination with BSC once daily for 3 weeks of continuous dosing followed by a 1-week break during a treatment cycle (Each cycle length was 28 days).
- Placebo + BSC Group: Participants received placebo matched to fruquintinib oral capsule in combination with BSC once daily for 3 weeks of continuous dosing followed by a 1-week break during a treatment cycle (Each cycle length was 28 days).
Period: Overall Study
Arm/Group | Fruquintinib + Best Supportive Care (BSC) Group | Placebo + BSC Group
Started | 461 | 230
Safety Population (SP) (The Safety population (SP) included all randomized participants who received at least 1 dose of study drug.) | 456 | 230
Pharmacokinetic (PK) Population (The Pharmacokinetic (PK) population included all participants who received at least 1 dose of study drug and had at least 1 post dose PK sample collected and analyzed.) | 329 | 2
Completed | 0 | 0
Not Completed | 461 | 230
Not completed — Adverse Event | 2 | 0
Not completed — Death | 411 | 203
Not completed — Lost to Follow-up | 3 | 1
Not completed — Withdrawal of consent | 14 | 8
Not completed — Radiological Disease Progression | 6 | 0
Not completed — Sponsor Decision | 19 | 14
Not completed — Other | 6 | 4

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) population included all randomized participants.
Groups:
- Fruquintinib + BSC Group: Participants received 5 mg of fruquintinib oral capsule in combination with BSC once daily for 3 weeks of continuous dosing followed by a 1-week break during a treatment cycle (Each cycle length was 28 days).
- Total: Total of all reporting groups
Arm/Group | Fruquintinib + BSC Group | Placebo + BSC Group | Total
Number analyzed (Participants) | 461 | 230 | 691
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.2 (10.41) | 62.4 (9.67) | 62.2 (10.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 216 | 90 | 306
  Male | 245 | 140 | 385
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 14 | 34
  Not Hispanic or Latino | 405 | 202 | 607
  Unknown or Not Reported | 36 | 14 | 50
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0 | 1 | 1
  Race: Asian | 43 | 18 | 61
  Race: Black or African American | 13 | 7 | 20
  Race: Native Hawaiian or Other | 3 | 2 | 5
  Race: White | 367 | 192 | 559
  Race: Other | 5 | 2 | 7
  Race: Multiple races | 2 | 0 | 2
  Race: Not reported/unknown | 28 | 8 | 36

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the time (months) from date of randomization to death from any cause. OS was calculated as (date of death or last known alive - date of randomization + 1)/30.4375. Participants without report of death at the time of analysis will be censored at the date last known alive.
Time Frame: From date of randomization to death from any cause (up to 22 months)
Population: ITT population included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Fruquintinib + BSC Group | Placebo + BSC Group
Number analyzed (Participants) | 461 | 230
months | 7.4 [6.7 to 8.2] | 4.8 [4.0 to 5.8]
Statistical Analysis 1: Comparison: Fruquintinib + BSC Group vs Placebo + BSC Group; Test type: Superiority; p < .001, stratified log-rank test — Raw unadjusted p-value was obtained by using a stratified log-rank test accounting for the randomization schedule stratification factors; Stratified Hazard Ratio = 0.662, 95% CI 2-sided [0.549 to 0.800] — The HR between 2 treatment groups (fruquintinib vs placebo), together with its 95 percent (%) confidence interval (CI), was calculated from a stratified Cox proportional hazards model accounting for the randomization schedule stratification factors

2. Secondary Outcome: Progression Free Survival (PFS), as Assessed by the Investigator Using Response Evaluation Criteria In Solid Tumors (RECIST) v1.1
Description: PFS was defined as the time (months) from randomization until the first radiographic documentation of objective progression as assessed by investigator using RECIST v1.1, or death from any cause, whichever comes first. More specifically, PFS was determined using all data until the last evaluable visit prior to or on the date of: (i) radiographic disease progression (PD) per RECIST v1.1; (ii) withdrawal of consent to obtain additional scans on study; or (iii) initiation of subsequent anticancer therapy other than the study drugs, whichever was earlier. PD was defined as: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study, including baseline; an absolute increase of at least 5 mm in the sum of diameters of target lesions; and the appearance of one or more new lesions.
Time Frame: From randomization until the first documentation of objective progression or death, whichever comes first (up to 22 months)
Population: ITT population included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Fruquintinib + BSC Group | Placebo + BSC Group
Number analyzed (Participants) | 461 | 230
months | 3.7 [3.5 to 3.8] | 1.8 [1.8 to 1.9]
Statistical Analysis 1: Comparison: Fruquintinib + BSC Group vs Placebo + BSC Group; Test type: Superiority; p < .001, stratified log-rank test — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.321, 95% CI 2-sided [0.267 to 0.386] — The HR between the 2 treatment groups (fruquintinib vs placebo), together with its 95% CI, was calculated from a stratified Cox proportional hazards model accounting for the randomization schedule stratification factors

3. Secondary Outcome: Objective Response Rate (ORR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Description: ORR was defined as the percentage of participants who achieved a best overall response of confirmed complete response (CR) or partial response (PR), per RECIST v1.1, as determined by the investigator. PR: At least a 30 percent (%) decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<)10 millimeters (mm).
Time Frame: From randomization until the first documentation of best overall response (up to 22 months)
Population: ITT population included all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fruquintinib + BSC Group | Placebo + BSC Group
Number analyzed (Participants) | 461 | 230
percentage of participants | 1.5 [0.6 to 3.1] | 0 [0.0 to 1.6]
Statistical Analysis 1: Comparison: Fruquintinib + BSC Group vs Placebo + BSC Group; Test type: Superiority; p = .059, Cochran-Mantel-Haenszel — p-value was calculated from a stratified Cochran-Mantel Haenszel test accounting for the randomization schedule stratification factors; Adjusted difference = 1.5, 95% CI 2-sided [0.4 to 2.7] — The adjusted difference and its 95% CI were calculated using the Wald method from Cochran-Mantel Haenszel test to account for the randomization schedule stratification factors

4. Secondary Outcome: Disease Control Rate (DCR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Description: DCR was defined as percentage of participants achieving a best overall response of confirmed CR, PR, or stable disease (SD) (for at least 7 weeks) per RECIST v1.1, as determined by the investigator. PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum on study. PD: At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (nadir), including baseline.
Time Frame: From randomization until the first documentation of best overall response (up to 22 months)
Population: ITT population included all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fruquintinib + BSC Group | Placebo + BSC Group
Number analyzed (Participants) | 461 | 230
percentage of participants | 55.5 [50.9 to 60.1] | 16.1 [11.6 to 21.5]
Statistical Analysis 1: Comparison: Fruquintinib + BSC Group vs Placebo + BSC Group; Test type: Superiority; p < .001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Adjusted difference = 39.4, 95% CI 2-sided [32.8 to 46.0] — [estimate comment as in outcome 3, analysis 1]

5. Secondary Outcome: Duration of Response (DOR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Description: DOR was defined as the time (in months) from the first occurrence of PR or CR by RECIST Version 1.1, until the first date that progressive disease is documented by RECIST Version 1.1, or death, whichever comes first. Only those participants with confirmed responses of CR or PR were included in this analysis. DOR was calculated as (date of death or PD or last assessment - date of first occurrence of confirmed CR or PR + 1)/30.4375.
Time Frame: From first occurrence of PR or CR until the first documentation progression or death, whichever comes first (up to 22 months
Population: Analysis was performed on subset of participants who had a response. Here, '0' in 'overall number of participants analyzed represents that DOR could only be analyzed in participants who achieved a response. As no participant in the Placebo Plus BSC Group cohort achieved any response, no DOR is available.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Fruquintinib + BSC Group | Placebo + BSC Group
Number analyzed (Participants) | 7 | 0
months | 10.7 [3.9 to NA] — Upper limit of 95% CI was not estimable due to limited number of participants with events. |

6. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An adverse event (AE) was any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE was considered a TEAE if the onset date was on or after the start of study treatment or if the onset date was missing, or if the AE had an onset date before the start of study treatment but worsened in severity after the study treatment until 30 days after the last dose of study treatment or a new treatment of anti-tumor therapy, whichever was earlier. After this period, treatment-related SAEs were also considered as TEAEs. AEs with an unknown/not reported onset date were also included.
Time Frame: From start of study drug administration up to approximately 40 months
Population: SP included all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Fruquintinib + BSC Group | Placebo + BSC Group
Number analyzed (Participants) | 456 | 230
Participants
  Participants with TEAEs | 451 | 214
  Participants with Serious TEAEs | 173 | 88

7. Secondary Outcome: Observed Plasma Concentrations of Fruquintinib and Metabolite M11
Description: Plasma samples were collected from the participants at the defined time points. Plasma concentrations were measured using a validated, specific, and sensitive liquid chromatography tandem mass spectrometry method. M11 is the active metabolite for the study drug.
Time Frame: Cycle 1 (Day 1 and 21): Pre-dose, 1, 2, 3 and 4 hours; Cycle 2 (Day 21): Predose and 2 hours, Cycle 3 (Day 1): Pre-dose, Cycle 3 (Day 21): Pre-dose and 2 hours, Cycle 5, 7, 9, 11, 13, 15 and 17 (Day 1): Pre-dose (Each cycle = 28 days)
Population: PK population was used for tabulation of fruquintinib and M11 concentrations from PK plasma samples collected from the Fruquintinib + BSC Group. PK samples for the Placebo + BSC Group were not analyzed. Here, "Overall Number of Participants Analyzed" signifies those participants in the Fruquintinib + BSC Group who were evaluable for this outcome measure and "number analyzed" signifies those participants who were evaluable at the specified timepoints.
Measure: Mean (Standard Deviation); unit: nanogram/milliliter (ng/mL)
Arm/Group | Fruquintinib + BSC Group
Number analyzed (Participants) | 312
nanogram/milliliter (ng/mL)
  Cycle 1 Day 1 - Pre-dose (Plasma Concentrations of Fruquintinib) | 2.90 (19.9)
  Cycle 1 Day 1 - Pre-dose (Plasma Concentrations of M11) | 0.585 (6.61)
  Cycle 1 Day 1 - 1 hour (Plasma Concentrations of Fruquintinib): number analyzed (Participants) | 171
  Cycle 1 Day 1 - 1 hour (Plasma Concentrations of Fruquintinib) | 59.9 (51.0)
  Cycle 1 Day 1 - 1 hour (Plasma Concentrations of M11): number analyzed (Participants) | 171
  Cycle 1 Day 1 - 1 hour (Plasma Concentrations of M11) | 1.06 (8.36)
  Cycle 1 Day 1 - 2 hours (Plasma Concentrations of Fruquintinib): number analyzed (Participants) | 304
  Cycle 1 Day 1 - 2 hours (Plasma Concentrations of Fruquintinib) | 91.5 (48.2)
  Cycle 1 Day 1 - 2 hours (Plasma Concentrations of M11): number analyzed (Participants) | 304
  Cycle 1 Day 1 - 2 hours (Plasma Concentrations of M11) | 1.03 (6.81)
  Cycle 1 Day 1 - 3 hours (Plasma Concentrations of Fruquintinib): number analyzed (Participants) | 171
  Cycle 1 Day 1 - 3 hours (Plasma Concentrations of Fruquintinib) | 98.5 (47.1)
  Cycle 1 Day 1 - 3 hours (Plasma Concentrations of M11): number analyzed (Participants) | 171
  Cycle 1 Day 1 - 3 hours (Plasma Concentrations of M11) | 1.96 (9.51)
  Cycle 1 Day 1 - 4 hours (Plasma Concentrations of Fruquintinib): number analyzed (Participants) | 171
  Cycle 1 Day 1 - 4 hours (Plasma Concentrations of Fruquintinib) | 99.7 (44.6)
  Cycle 1 Day 1 - 4 hours (Plasma Concentrations of M11): number analyzed (Participants) | 171
  Cycle 1 Day 1 - 4 hours (Plasma Concentrations of M11) | 2.71 (10.7)
  Cycle 1 Day 21 - Pre-dose (Plasma Concentrations of Fruquintinib): number analyzed (Participants) | 227
  Cycle 1 Day 21 - Pre-dose (Plasma Concentrations of Fruquintinib) | 219 (82.6)
  Cycle 1 Day 21 - Pre-dose (Plasma Concentrations of M11): number analyzed (Participants) | 227
  Cycle 1 Day 21 - Pre-dose (Plasma Concentrations of M11) | 94.5 (52.6)
  Cycle 1 Day 21 - 1 hour (Plasma Concentrations of Fruquintinib): number analyzed (Participants) | 112
  Cycle 1 Day 21 - 1 hour (Plasma Concentrations of Fruquintinib) | 255 (101)
  Cycle 1 Day 21 - 1 hour (Plasma Concentrations of M11): number analyzed (Participants) | 112
  Cycle 1 Day 21 - 1 hour (Plasma Concentrations of M11) | 92.0 (54.3)
  Cycle 1 Day 21 - 2 hours (Plasma Concentrations of Fruquintinib): number analyzed (Participants) | 214
  Cycle 1 Day 21 - 2 hours (Plasma Concentrations of Fruquintinib) | 279 (91.6)
  Cycle 1 Day 21 - 2 hours (Plasma Concentrations of M11): number analyzed (Participants) | 214
  Cycle 1 Day 21 - 2 hours (Plasma Concentrations of M11) | 89.9 (49.5)
  Cycle 1 Day 21 -3 hours (Plasma Concentrations of Fruquintinib): number analyzed (Participants) | 113
  Cycle 1 Day 21 -3 hours (Plasma Concentrations of Fruquintinib) | 293 (95.2)
  Cycle 1 Day 21 - 3 hours (Plasma Concentrations of M11): number analyzed (Participants) | 113
  Cycle 1 Day 21 - 3 hours (Plasma Concentrations of M11) | 88.0 (50.4)
  Cycle 1 Day 21 - 4 hours (Plasma Concentrations of Fruquintinib): number analyzed (Participants) | 114
  Cycle 1 Day 21 - 4 hours (Plasma Concentrations of Fruquintinib) | 294 (88.0)
  Cycle 1 Day 21 - 4 hours (Plasma Concentrations of M11): number analyzed (Participants) | 114
  Cycle 1 Day 21 - 4 hours (Plasma Concentrations of M11) | 89.2 (49.0)
  Cycle 2 Day 21 - Predose (Plasma Concentrations of Fruquintinib): number analyzed (Participants) | 204
  Cycle 2 Day 21 - Predose (Plasma Concentrations of Fruquintinib) | 222 (82.0)
  Cycle 2 Day 21 - Predose (Plasma Concentrations of M11): number analyzed (Participants) | 204
  Cycle 2 Day 21 - Predose (Plasma Concentrations of M11) | 97.6 (53.7)
  Cycle 2 Day 21 - 2 hours (Plasma Concentrations of Fruquintinib): number analyzed (Participants) | 193
  Cycle 2 Day 21 - 2 hours (Plasma Concentrations of Fruquintinib) | 284 (95.2)
  Cycle 2 Day 21 - 2 hours (Plasma Concentrations of M11): number analyzed (Participants) | 193
  Cycle 2 Day 21 - 2 hours (Plasma Concentrations of M11) | 94.2 (52.8)
  Cycle 3 Day 1 - Pre-dose (Plasma Concentrations of Fruquintinib): number analyzed (Participants) | 177
  Cycle 3 Day 1 - Pre-dose (Plasma Concentrations of Fruquintinib) | 16.7 (18.9)
  Cycle 3 Day 1 - Pre-dose (Plasma Concentrations of M11): number analyzed (Participants) | 177
  Cycle 3 Day 1 - Pre-dose (Plasma Concentrations of M11) | 22.6 (18.2)
  Cycle 3 Day 21 - Pre-dose (Plasma Concentrations of Fruquintinib): number analyzed (Participants) | 137
  Cycle 3 Day 21 - Pre-dose (Plasma Concentrations of Fruquintinib) | 212 (74.6)
  Cycle 3 Day 21 - Pre-dose (Plasma Concentrations of M11): number analyzed (Participants) | 137
  Cycle 3 Day 21 - Pre-dose (Plasma Concentrations of M11) | 90.6 (54.1)
  Cycle 3 Day 21 - 2 hours (Plasma Concentrations of Fruquintinib): number analyzed (Participants) | 123
  Cycle 3 Day 21 - 2 hours (Plasma Concentrations of Fruquintinib) | 275 (78.6)
  Cycle 3 Day 21 - 2 hours (Plasma Concentrations of M11): number analyzed (Participants) | 123
  Cycle 3 Day 21 - 2 hours (Plasma Concentrations of M11) | 92.8 (54.2)
  Cycle 5 Day 1 - Pre-Dose (Plasma Concentrations of Fruquintinib): number analyzed (Participants) | 103
  Cycle 5 Day 1 - Pre-Dose (Plasma Concentrations of Fruquintinib) | 16.9 (20.5)
  Cycle 5 Day 1 - Pre-Dose (Plasma Concentrations of M11): number analyzed (Participants) | 103
  Cycle 5 Day 1 - Pre-Dose (Plasma Concentrations of M11) | 23.2 (20.9)
  Cycle 7 Day 1 - Pre-Dose (Plasma Concentrations of Fruquintinib: number analyzed (Participants) | 46
  Cycle 7 Day 1 - Pre-Dose (Plasma Concentrations of Fruquintinib | 18.2 (33.0)
  Cycle 7 Day 1 - Pre-Dose (Plasma Concentrations of M11): number analyzed (Participants) | 46
  Cycle 7 Day 1 - Pre-Dose (Plasma Concentrations of M11) | 20.1 (12.1)
  Cycle 9 Day 1 - Pre-Dose (Plasma Concentrations of Fruquintinib): number analyzed (Participants) | 13
  Cycle 9 Day 1 - Pre-Dose (Plasma Concentrations of Fruquintinib) | 12.2 (12.6)
  Cycle 9 Day 1 - Pre-Dose (Plasma Concentrations of M11): number analyzed (Participants) | 13
  Cycle 9 Day 1 - Pre-Dose (Plasma Concentrations of M11) | 19.1 (17.1)
  Cycle 11 Day 1 - Pre-Dose (Plasma Concentrations of Fruquintinib): number analyzed (Participants) | 6
  Cycle 11 Day 1 - Pre-Dose (Plasma Concentrations of Fruquintinib) | 13.4 (13.4)
  Cycle 11 Day 1 - Pre-Dose (Plasma Concentrations of M11): number analyzed (Participants) | 6
  Cycle 11 Day 1 - Pre-Dose (Plasma Concentrations of M11) | 17.1 (15.3)
  Cycle 13 Day 1 - Pre-Dose (Plasma Concentrations of Fruquintinib): number analyzed (Participants) | 1
  Cycle 13 Day 1 - Pre-Dose (Plasma Concentrations of Fruquintinib) | 15.4
  Cycle 13 Day 1 - Pre-Dose (Plasma Concentrations of M11): number analyzed (Participants) | 1
  Cycle 13 Day 1 - Pre-Dose (Plasma Concentrations of M11) | 23.1
  Cycle 15 Day 1 - Pre-Dose (Plasma Concentrations of Fruquintinib): number analyzed (Participants) | 1
  Cycle 15 Day 1 - Pre-Dose (Plasma Concentrations of Fruquintinib) | 10.8
  Cycle 15 Day 1 - Pre-Dose (Plasma Concentrations of M11): number analyzed (Participants) | 1
  Cycle 15 Day 1 - Pre-Dose (Plasma Concentrations of M11) | 19.2
  Cycle 17 Day 1 - Pre-Dose (Plasma Concentrations of Fruquintinib): number analyzed (Participants) | 1
  Cycle 17 Day 1 - Pre-Dose (Plasma Concentrations of Fruquintinib) | 10.6
  Cycle 17 Day 1 - Pre-Dose (Plasma Concentrations of M11): number analyzed (Participants) | 1
  Cycle 17 Day 1 - Pre-Dose (Plasma Concentrations of M11) | 15.2

8. Secondary Outcome: Change From Baseline of Electrocardiogram (ECG) Results - QTcF Intervals Using Fridericia's Formula
Description: QT Interval: Ventricular depolarization plus ventricular repolarization Normal Range: 400 to 460 milliseconds (msec). QTc: QT interval corrected based on the patient's heart rate. QTcF: An electrocardiographic finding in which the QT interval corrected for heart rate using Fridericia's formula. QTc = QT/∛(RR) RR = Respiration rate.
Time Frame: Baseline, Cycle 1 (Day 1 and 21): Pre-dose, 1, 2, 3 and 4 hours; Cycle 2 and 3 (Day 21): Pre-dose (Each cycle = 28 days)
Population: SP included all randomized participants who received at least 1 dose of study drug. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure and "number analyzed" signifies those participants who were evaluable at the specified time points.
Measure: Mean (Standard Deviation); unit: millisecond (msec)
Arm/Group | Fruquintinib + BSC Group | Placebo + BSC Group
Number analyzed (Participants) | 272 | 131
millisecond (msec)
  Cycle 1 Day 1 - Pre-dose: number analyzed (Participants) | 261 | 126
  Cycle 1 Day 1 - Pre-dose | 1.9 (21.33) | 0.1 (17.95)
  Cycle 1 Day 1 - 1 hour: number analyzed (Participants) | 149 | 71
  Cycle 1 Day 1 - 1 hour | -0.1 (19.60) | 2.5 (19.70)
  Cycle 1 Day 1 - 2 hours | 1.9 (22.58) | 3.5 (20.13)
  Cycle 1 Day 1 - 3 hours: number analyzed (Participants) | 143 | 70
  Cycle 1 Day 1 - 3 hours | 2.6 (19.77) | 3.3 (18.03)
  Cycle 1 Day 1 - 4 hours: number analyzed (Participants) | 136 | 67
  Cycle 1 Day 1 - 4 hours | 1.2 (20.48) | 0.9 (17.66)
  Cycle 1 Day 21 - Pre-dose: number analyzed (Participants) | 184 | 95
  Cycle 1 Day 21 - Pre-dose | 3.2 (20.94) | -2.2 (20.31)
  Cycle 1 Day 21 - 1 hour: number analyzed (Participants) | 109 | 62
  Cycle 1 Day 21 - 1 hour | 4.0 (19.56) | -0.2 (16.77)
  Cycle 1 Day 21 - 2 hours: number analyzed (Participants) | 222 | 121
  Cycle 1 Day 21 - 2 hours | 5.0 (20.06) | 2.8 (18.23)
  Cycle 1 Day 21 - 3 hours: number analyzed (Participants) | 111 | 61
  Cycle 1 Day 21 - 3 hours | 5.9 (19.46) | 0.2 (14.70)
  Cycle 1 Day 21 - 4 hours: number analyzed (Participants) | 103 | 58
  Cycle 1 Day 21 - 4 hours | 3.9 (20.98) | -0.6 (18.13)
  Cycle 2 Day 21 - 2 hours: number analyzed (Participants) | 229 | 86
  Cycle 2 Day 21 - 2 hours | 1.4 (22.41) | 4.9 (24.28)
  Cycle 3 Day 21 - 2 hours: number analyzed (Participants) | 141 | 28
  Cycle 3 Day 21 - 2 hours | 2.6 (31.61) | 2.0 (20.08)

9. Secondary Outcome: Change From Baseline of ECG Results -QTcB Intervals Using Bazzett's Formula
Description: QT Interval: Ventricular depolarization plus ventricular repolarization Normal Range: 400 to 460 msec. QTc: QT interval corrected based on the patient's heart rate. QTcB: An electrocardiographic finding in which the QT interval corrected for heart rate using Bazzett's formula.
Time Frame: as for outcome 8
Population: SP included all randomized participants who received at least 1 dose of study drug. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure and "Number analyzed" signifies those participants who were evaluable at the specified timepoints.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Fruquintinib + BSC Group | Placebo + BSC Group
Number analyzed (Participants) | 258 | 122
msec
  Cycle 1 Day 1 - Pre-dose: number analyzed (Participants) | 249 | 118
  Cycle 1 Day 1 - Pre-dose | 2.9 (39.49) | 0.3 (20.55)
  Cycle 1 Day 1 - 1 hour: number analyzed (Participants) | 142 | 69
  Cycle 1 Day 1 - 1 hour | -3.1 (23.95) | 1.9 (20.11)
  Cycle 1 Day 1 - 2 hours | -2.0 (23.95) | 1.9 (20.11)
  Cycle 1 Day 1 - 3 hours: number analyzed (Participants) | 136 | 68
  Cycle 1 Day 1 - 3 hours | -0.9 (24.47) | 3.9 (19.75)
  Cycle 1 Day 1 - 4 hours: number analyzed (Participants) | 130 | 65
  Cycle 1 Day 1 - 4 hours | -1.9 (24.47) | 2.4 (20.11)
  Cycle 1 Day 21 - Pre-dose: number analyzed (Participants) | 177 | 91
  Cycle 1 Day 21 - Pre-dose | 3.9 (49.99) | 5.0 (50.43)
  Cycle 1 Day 21 - 1 hour: number analyzed (Participants) | 177 | 60
  Cycle 1 Day 21 - 1 hour | -1.3 (25.60) | 0.9 (20.48)
  Cycle 1 Day 21 - 2 hours: number analyzed (Participants) | 212 | 117
  Cycle 1 Day 21 - 2 hours | 1.6 (42.28) | 4.3 (19.57)
  Cycle 1 Day 21 - 3 hours: number analyzed (Participants) | 107 | 59
  Cycle 1 Day 21 - 3 hours | 1.2 (25.41) | 2.9 (18.29)
  Cycle 1 Day 21 - 4 hours: number analyzed (Participants) | 99 | 56
  Cycle 1 Day 21 - 4 hours | 0.2 (25.91) | 2.8 (20.13)
  Cycle 2 Day 21 - 2 hours: number analyzed (Participants) | 213 | 83
  Cycle 2 Day 21 - 2 hours | 1.7 (40.61) | 5.9 (24.96)
  Cycle 3 Day 21 - 2 hours: number analyzed (Participants) | 132 | 28
  Cycle 3 Day 21 - 2 hours | 4.2 (72.35) | 1.6 (22.06)

10. Secondary Outcome: Correlation Between Fruquintinib Exposure (CminSS) and Efficacy Parameters (OS)
Description: Model-predicted steady-state minimum plasma concentrations (CminSS) of fruquintinib based on the starting dose or adjusted for relative dose intensity [RDI] were used as the exposure measures in the efficacy exposure-response analyses. The correlation between OS and exposure was estimated using multivariable Cox proportional hazards modeling. OS was analyzed as time-to-event variable using a survival model. The efficacy exposure-response analyses included participants with mCRC and pooled the data from the fruquintinib group of current Study 2019-013-GLOB1 (N=328) and from Cohort B of Study 2015-013-00US1 (NCT03251378) (N=40) as per planned analysis. Here, the "unit of measure" i.e., '1/(nanogram per milliliter [ng/mL])', corresponds to the coefficient that describes the relationship between the probability of survival and CminSS value.
Time Frame: Up to 22 months
Population: The efficacy exposure-response analyses included participants who were evaluable for the population PK analysis and therefore had PK parameter estimates to enable estimation of fruquintinib exposure and evaluated for the parameter/endpoint in question. Here, "overall number of participants analyzed" signified those participants who were evaluable for this outcome measure. The population for this measure included participants from both studies 2015-013-00US1 and the current study.
Measure: Number; unit: 1/(ng/mL)
Groups:
- Fruquintinib: Pooled Studies for Exposure and Efficacy Analysis: Participants in the current 2019-013-GLOB1 (NCT04322539) study received 5 mg of fruquintinib oral capsules with BSC once daily for 3 weeks of continuous dosing, followed by a 1-week break during each 28-day treatment cycle. Participants in Cohort B of Study 2015-013-00US1 (NCT03251378) with metastatic colorectal carcinoma (mCRC) and treatment with chemotherapy and trifluridine, tipiracil, and/or regorafenib received fruquintinib 5 mg capsules, once daily, for 3 weeks on and 1 week off in each 28-day treatment cycle until disease progression, unacceptable toxicity, use of other antitumor treatment, withdrawal of consent, or discontinuation by the Investigator, whichever occurred first.
Arm/Group | Fruquintinib: Pooled Studies for Exposure and Efficacy Analysis
Number analyzed (Participants) | 368
1/(ng/mL)
  CminSS Coefficient Based on the Starting Dose for OS Exposure-Response Analyses | 0.00193
  CminSS Coefficient Based on the Adjusted RDI for OS Exposure-Response Analyses | 0.000407
Statistical Analysis 1: Comparison: Fruquintinib: Pooled Studies for Exposure and Efficacy Analysis; CminSS Based on the Starting Dose for OS Exposure-Response Analyses; Test type: Other; p = 0.0600, Wald test
Statistical Analysis 2: Comparison: Fruquintinib: Pooled Studies for Exposure and Efficacy Analysis; CminSS Based on the Adjusted RDI for OS Exposure-Response Analyses; Test type: Other; p = 0.8065, Wald test

11. Secondary Outcome: Correlation Between Fruquintinib Exposure (CmaxSS) and Safety Parameters (Any Grade [Gr] and Grade 3+ (Gr3+): Dermatological Toxicity, Proteinuria and Gr Hemorrhage)
Description: Model-predicted steady-state maximum plasma concentration (CmaxSS) of fruquintinib based on the assigned dose of fruquintinib were investigated as fruquintinib exposure measure for the safety exposure-response analyses. The correlation between exposure and the probability of experiencing these AEs was evaluated using logistic regression analysis, with the slope serving as the estimate. The safety exposure-response analysis included participants with cancer, and the data of this outcome measure were pooled with data from the following studies as per the planned analysis: 2019-013-GLOB1 (NCT04322539) (N=334), 2009-013-00CH1 (NCT01645215) (N=40), 2012-013-00CH3 (NCT01975077) (N=40), and 2015-013-00US1 (NCT03251378) (N=101). Here, the "unit of measure" i.e., '1/(ng/mL)', corresponds to the coefficient that describes the relationship between the probability of occurrence of the safety parameter and CmaxSS value.
Time Frame: Up to 22 months
Population: Safety exposure-response analyses included participants who were evaluable for population PK analysis and therefore had PK parameter estimates to enable estimation of fruquintinib exposure and evaluated for parameter/endpoint in question. Here, "overall number of participants analyzed" signified those participants who were evaluable for this outcome measure. The population for this measure included participants from 2019-013-GLOB1, 2009-013-00CH1, 2012-013-00CH3, and 2015-013-00US1.
Measure: Number; unit: 1/(ng/mL)
Groups:
- Fruquintinib: Pooled Studies for Exposure and Safety Analysis: Participants in the current 2019-013-GLOB1 (NCT04322539) study received 5 mg of fruquintinib oral capsules once daily for 3 weeks of continuous dosing, followed by a 1-week break during each 28-day treatment cycle. Participants in the 2009-013-00CH1 (NCT01645215) study received 1 mg to 6 mg of fruquintinib oral capsule once daily and 5 mg to 6 mg of fruquintinib oral capsule for 3 weeks on and 1 week off during each 28-day treatment cycle. Participants in the 2012-013-00CH3 (NCT01975077) study received 4 mg of fruquintinib capsule once daily in 28-day cycles. Participants in the Study 2015-013-00US1 (NCT03251378) with advanced solid tumors of any type or with mCRC received fruquintinib 3 mg or 5 mg once daily for 3 weeks on and 1 week off in each 28-day treatment cycle until disease progression, unacceptable toxicity, use of other antitumor treatment, withdrawal of consent, or discontinuation by the Investigator, whichever occurred first.
Arm/Group | Fruquintinib: Pooled Studies for Exposure and Safety Analysis
Number analyzed (Participants) | 515
1/(ng/mL)
  CmaxSS Coefficient for Gr Dermatological toxicity for Exposure-Response Analyses | 0.00134
  CmaxSS Coefficient for Gr3+ Dermatological Toxicity for Exposure-Response Analyses | 0.00411
  CmaxSS Coefficient for Gr Proteinuria for Exposure-Response Analyses | -0.00101
  CmaxSS Coefficient for Gr3+ Proteinuria for Exposure-Response Analyses | 0.00143
  CmaxSS Coefficient for Gr Hemorrhage for Exposure-Response Analyses | 0.00180
Statistical Analysis 1: Comparison: Fruquintinib: Pooled Studies for Exposure and Safety Analysis; CmaxSS for Gr Dermatological toxicity for Exposure-Response Analyses; Test type: Other; p = 0.265, Wald test
Statistical Analysis 2: Comparison: Fruquintinib: Pooled Studies for Exposure and Safety Analysis; CmaxSS for Gr3+ Dermatological Toxicity for Exposure-Response Analyses; Test type: Other; p = 0.0159, Wald test
Statistical Analysis 3: Comparison: Fruquintinib: Pooled Studies for Exposure and Safety Analysis; CmaxSS for Gr Proteinuria for Exposure-Response Analyses; Test type: Other; p = 0.484, Wald test
Statistical Analysis 4: Comparison: Fruquintinib: Pooled Studies for Exposure and Safety Analysis; CmaxSS for Gr3+ Proteinuria for Exposure-Response Analyses; Test type: Other; p = 0.642, Wald test
Statistical Analysis 5: Comparison: Fruquintinib: Pooled Studies for Exposure and Safety Analysis; CmaxSS for Gr Hemorrhage for Exposure-Response Analyses; Test type: Other; p = 0.166, Wald test

12. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life (QOL) Questionnaire Core 30 (EORTC QLQ-C30) Global Health Status/Quality of Life Scale Score
Description: EORTC QLQ-C30 contains 30 items across 5 functional scales (physical, role, cognitive, emotional, and social), 9 symptom scales (fatigue, nausea and vomiting, pain, dyspnea, sleep disturbance, appetite loss, constipation, diarrhea, and financial difficulties) and global health status/QOL scale. EORTC QLQ-C30 contains 28 questions (4-point scale where 1=Not at all [best] to 4=Very Much [worst]) and 2 questions (7-point scale where 1=Very poor [worst] to 7= Excellent [best]). Raw scores are standardized and converted into scale scores ranging from 0 to 100. For global health status/QOL scale, higher scores represent better QOL. A negative change from baseline value indicates patient condition worsened. Change from baseline in the EORTC QLQ-C30 Global Health Status/Quality of Life Scale scores was performed by visit (i.e., cycle), using a restricted maximum likelihood (REML)-based mixed model repeated measures (MMRM) approach.
Time Frame: Baseline, Cycle 2, 3 and 4 (Each cycle=28 days)
Population: ITT population included all randomized participants. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure and "Number analyzed" signifies those participants who were evaluable at the specified timepoints.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Fruquintinib + BSC Group | Placebo + BSC Group
Number analyzed (Participants) | 330 | 149
score on a scale
  Cycle 2 | -2.1 (1.59) | -3.7 (1.95)
  Cycle 3: number analyzed (Participants) | 229 | 53
  Cycle 3 | -4.5 (1.69) | -6.1 (2.54)
  Cycle 4: number analyzed (Participants) | 182 | 29
  Cycle 4 | -4.2 (1.76) | -2.1 (3.03)

13. Secondary Outcome: Change From Baseline in EuroQoL 5 Dimension 5 Level (EQ-5D-5L) Visual Analog Scale (VAS) Score
Description: The EQ-5D-5L is a self-reported health status questionnaire that consisted of six questions used to calculate a health utility score. There were two components to the EQ-5D-5L: a five-item health state profile that assessed mobility, self-care, usual activities, pain/discomfort, and anxiety/depression used to obtain an Index Utility Score and a general VAS score for health status. EQ-5D VAS was used to record participant's rating for his/her current health-related quality of life state on a vertical VAS with scores ranging from 0 to 100, where 0 = worst imaginable health state and 100 = best imaginable health state. The higher the score the better the health status. A negative change from baseline value represents patient condition worsened. Change from baseline in the EQ-5D-5L VAS scores was performed by visit (i.e. cycle), using a REML-based MMRM approach.
Time Frame: Baseline, Cycle 2, 3 and 4 (Each cycle=28 days)
Population: ITT population included all randomized participants. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure and "Number analyzed" signifies those participants who were evaluable at the specified categories.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Fruquintinib + BSC Group | Placebo + BSC Group
Number analyzed (Participants) | 388 | 230
score on a scale
  Cycle 2: number analyzed (Participants) | 337 | 151
  Cycle 2 | -0.3 (1.38) | -0.9 (1.69)
  Cycle 3: number analyzed (Participants) | 232 | 54
  Cycle 3 | -1.1 (1.48) | -2.5 (2.22)
  Cycle 4: number analyzed (Participants) | 185 | 30
  Cycle 4 | -4.0 (1.59) | -2.1 (2.79)

14. Secondary Outcome: Change From Baseline in EuroQoL 5 Dimension 5 Level (EQ-5D-5L) Health Utility Index Scores
Description: EQ-5D-5L consisted of 2 components: health state profile and optional VAS. EQ-5D health state profile had 5 dimensions: mobility, self-care, usual activities, pain/discomfort, anxiety/depression. Each dimension has 5 levels: 1= no problem, 2= slight problem, 3= moderate problem, 4= severe problem, and 5= extreme problem. The response levels collected from the EQ-5D-5L five dimensions as a health profile are converted into an EQ-5D-5L index (utility) scores to represent participants' utility value. The range of health utility index score is from -0.285 to 1, where higher value indicates perfect health and a negative value represents a state worse than dead. Change from baseline in EQ-5D-5L health utility index scores was performed by visit (i.e., cycle), using a REML-based MMRM approach.
Time Frame: Baseline, Cycle 2, 3 and 4 (Each cycle=28 days)
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Fruquintinib + BSC Group | Placebo + BSC Group
Number analyzed (Participants) | 337 | 151
score on a scale
  Cycle 2 | 0.0 (0.01) | 0.0 (0.02)
  Cycle 3: number analyzed (Participants) | 232 | 54
  Cycle 3 | 0.0 (0.01) | 0.0 (0.02)
  Cycle 4: number analyzed (Participants) | 185 | 30
  Cycle 4 | -0.1 (0.02) | 0.0 (0.03)

15. Secondary Outcome: Health Care Resource Utilization: Duration of Hospital Visits by Participants
Description: Duration of hospital visit was calculated as = stop date - start date + 1. Mean and standard deviation data for duration of hospital visits (in days) by participants was reported in this outcome measure.
Time Frame: From start of study drug administration up to 22 months
Population: ITT population included all randomized participants.
Measure: Mean (Standard Deviation); unit: days per visit
Units Other Than Participants: Number of visits
Arm/Group | Fruquintinib + BSC Group | Placebo + BSC Group
Number analyzed (Participants) | 461 | 230
Number analyzed (Number of visits) | 545 | 232
days per visit | 3.3 (6.81) | 4.4 (7.53)

16. Secondary Outcome: Health Care Resource Utilization: Number of Participants With Any Concomitant Medications Prescribed
Description: Number of participants with any concomitant medications prescribed were reported.
Time Frame: From start of study drug administration up to 22 months
Population: ITT population included all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Fruquintinib + BSC Group | Placebo + BSC Group
Number analyzed (Participants) | 461 | 230
Participants | 116 | 63

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to approximately 40 months
Description: All-Cause Mortality data collected during the study was assessed for all randomized participants. Serious AEs and Non-Serious AEs data were collected based on safety population that included all randomized participants who received at least 1 dose.
Arm/Group | Fruquintinib + BSC Group | Placebo + BSC Group
All-Cause Mortality (participants affected / at risk) | 411/461 | 203/230
Serious Adverse Events (participants affected / at risk) | 173/456 | 88/230
Other Adverse Events (participants affected / at risk) | 446/456 | 205/230
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fruquintinib + BSC Group (N=456) | Placebo + BSC Group (N=230)
Abdominal pain (Gastrointestinal disorders) | 7 | 2
Intestinal obstruction (Gastrointestinal disorders) | 7 | 6
Small intestinal obstruction (Gastrointestinal disorders) | 5 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 4 | 0
Constipation (Gastrointestinal disorders) | 3 | 0
Ileus (Gastrointestinal disorders) | 2 | 5
Intestinal perforation (Gastrointestinal disorders) | 4 | 0
Vomiting (Gastrointestinal disorders) | 3 | 3
Colitis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Small intestinal perforation (Gastrointestinal disorders) | 2 | 0
Stomatitis (Gastrointestinal disorders) | 2 | 1
Subileus (Gastrointestinal disorders) | 2 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Colonic fistula (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastric perforation (Gastrointestinal disorders) | 1 | 0
Gastrointestinal perforation (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Oesophageal obstruction (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Rectal perforation (Gastrointestinal disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 2
Ascites (Gastrointestinal disorders) | 0 | 1
Enterovesical fistula (Gastrointestinal disorders) | 0 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Rectal stenosis (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Disease progression (General disorders) | 27 | 28
General physical health deterioration (General disorders) | 10 | 5
Asthenia (General disorders) | 5 | 0
Pyrexia (General disorders) | 4 | 2
Condition aggravated (General disorders) | 3 | 2
Non-cardiac chest pain (General disorders) | 2 | 0
Chest pain (General disorders) | 1 | 0
Chills (General disorders) | 1 | 0
Death (General disorders) | 2 | 2
Discomfort (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 1
Ulcer (General disorders) | 1 | 0
Generalised oedema (General disorders) | 1 | 0
Pain (General disorders) | 0 | 1
Sudden death (General disorders) | 0 | 1
Pneumonia (Infections and infestations) | 9 | 1
Sepsis (Infections and infestations) | 5 | 0
Urinary tract infection (Infections and infestations) | 3 | 3
Abscess limb (Infections and infestations) | 1 | 0
Biliary tract infection (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 1 | 0
Empyema (Infections and infestations) | 1 | 1
Fournier's gangrene (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Perirectal abscess (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 1
COVID-19 (Infections and infestations) | 0 | 3
Coronavirus infection (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 1 | 1
Wound infection bacterial (Infections and infestations) | 0 | 1
Wound sepsis (Infections and infestations) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchopleural fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 5 | 1
Urinary tract obstruction (Renal and urinary disorders) | 3 | 0
Hydronephrosis (Renal and urinary disorders) | 2 | 0
Ureteric obstruction (Renal and urinary disorders) | 2 | 0
Haematuria (Renal and urinary disorders) | 1 | 1
Proteinuria (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 1
Vesicocutaneous fistula (Renal and urinary disorders) | 1 | 0
Biliary obstruction (Hepatobiliary disorders) | 3 | 1
Cholangitis (Hepatobiliary disorders) | 3 | 1
Hepatic failure (Hepatobiliary disorders) | 3 | 2
Cholecystitis (Hepatobiliary disorders) | 2 | 0
Bile duct stenosis (Hepatobiliary disorders) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 2
Hypertransaminasaemia (Hepatobiliary disorders) | 2 | 0
Jaundice (Hepatobiliary disorders) | 1 | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 2 | 0
Spinal cord compression (Nervous system disorders) | 2 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 1
Hepatic encephalopathy (Nervous system disorders) | 1 | 0
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 1
Fistula (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 6 | 0
Hypertensive crisis (Vascular disorders) | 2 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Haemorrhage (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 3 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0
Recall phenomenon (Injury, poisoning and procedural complications) | 1 | 0
Sternal fracture (Injury, poisoning and procedural complications) | 1 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour invasion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Blood bilirubin increased (Investigations) | 4 | 2
Blood creatinine increased (Investigations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Liver function test abnormal (Investigations) | 0 | 1
SARS-CoV-2 test positive (Investigations) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 2 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 2 | 1
Polycythaemia (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 2 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Female genital tract fistula (Reproductive system and breast disorders) | 1 | 0
Intermenstrual bleeding (Reproductive system and breast disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Device dislocation (Product Issues) | 1 | 0
Osteomyelitis chronic (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fruquintinib + BSC Group (N=456) | Placebo + BSC Group (N=230)
Asthenia (General disorders) | 153 | 52
Fatigue (General disorders) | 93 | 37
Mucosal inflammation (General disorders) | 62 | 6
Pyrexia (General disorders) | 43 | 22
Oedema peripheral (General disorders) | 23 | 17
Diarrhoea (Gastrointestinal disorders) | 113 | 24
Abdominal pain (Gastrointestinal disorders) | 80 | 36
Nausea (Gastrointestinal disorders) | 82 | 43
Constipation (Gastrointestinal disorders) | 75 | 22
Stomatitis (Gastrointestinal disorders) | 67 | 7
Vomiting (Gastrointestinal disorders) | 67 | 25
Abdominal pain upper (Gastrointestinal disorders) | 35 | 8
Hypertension (Vascular disorders) | 165 | 21
Weight decreased (Investigations) | 58 | 21
Aspartate aminotransferase increased (Investigations) | 50 | 10
Alanine aminotransferase increased (Investigations) | 49 | 8
Blood bilirubin increased (Investigations) | 33 | 10
Blood thyroid stimulating hormone increased (Investigations) | 32 | 3
Platelet count decreased (Investigations) | 28 | 2
Blood alkaline phosphatase increased (Investigations) | 24 | 10
Decreased appetite (Metabolism and nutrition disorders) | 127 | 41
Hypokalaemia (Metabolism and nutrition disorders) | 29 | 4
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 75 | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 39 | 21
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 39 | 22
Arthralgia (Musculoskeletal and connective tissue disorders) | 52 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 48 | 17
Pain in extremity (Musculoskeletal and connective tissue disorders) | 28 | 6
Hypothyroidism (Endocrine disorders) | 94 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 89 | 6
Proteinuria (Renal and urinary disorders) | 81 | 12
Anaemia (Blood and lymphatic system disorders) | 38 | 28
Thrombocytopenia (Blood and lymphatic system disorders) | 30 | 3
Headache (Nervous system disorders) | 40 | 10
Insomnia (Psychiatric disorders) | 26 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-21): https://cdn.clinicaltrials.gov/large-docs/39/NCT04322539/Prot_SAP_000.pdf